CLINICAL TRIAL: NCT01936688
Title: A 28-Week, Phase 3, Randomized, Active Comparator and Placebo-Controlled, Parallel Design Study to Evaluate the Efficacy and Safety/Tolerability of Subcutaneous SCH 900222 / MK-3222, Followed by an Optional Long-Term Safety Extension Study, in Subjects With Moderate-to-Severe Chronic Plaque Psoriasis (Protocol No. MK-3222-012)
Brief Title: A Study to Evaluate the Efficacy and Safety/Tolerability of Subcutaneous MK-3222 in Participants With Moderate-to-Severe Chronic Plaque Psoriasis (MK-3222-012)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3222-012; MK-3222-012 (Other: Merck Study Number); 2013-001740-54 (EudraCT Number)
Record Dates: First submitted 2013-09-03; First posted 2013-09-06 (Estimated); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Plaque-type Psoriasis
MeSH Terms: interventions — tildrakizumab; Etanercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- MK-3222 200 mg + Placebo to Etanercept (Experimental): MK-3222 200 mg subcutaneously (SC) on Weeks 0, 4, 16, and 28 and, optionally, every 12 weeks thereafter until Week 220, plus etanercept placebo twice weekly up to Week 12, and then once weekly through Week 28.
  Interventions: Drug: MK-3222 200 mg; Drug: Placebo to Etanercept
- MK-3222 100 mg + Placebo to Etanercept (Experimental): MK-3222 100 mg SC on Weeks 0, 4, 16, and 28 and, optionally, every 12 weeks thereafter until Week 220, plus etanercept placebo twice weekly up to Week 12, and then once weekly through Week 28.
  Interventions: Drug: MK-3222 100 mg; Drug: Placebo to Etanercept
- Placebo to MK-3222 + Placebo to Etanercept (Placebo Comparator): Placebo to MK-3222 administered SC on Weeks 0 and 4 plus etanercept placebo twice weekly up to Week 12, then once weekly up to Week 28. Participants will be re-randomized 1:1 at Week 12 to receive MK-3222 high dose or MK-3222 low dose on Weeks 12, 16, and 28 and, optionally, every 12 weeks thereafter through Week 220.
  Interventions: Drug: Placebo to MK-3222; Drug: Placebo to Etanercept
- Placebo to MK-3222 + Etanercept 50 mg (Active Comparator): Matching placebo to MK-3222 SC on Weeks 0 and 4 and etanercept 50 mg twice weekly up to Week 12 and then once weekly through Week 28.
  Interventions: Drug: Placebo to MK-3222; Drug: Etanercept 50 mg

INTERVENTIONS:
Drug: MK-3222 200 mg — MK-3222 200 mg administered SC.
  Arms: MK-3222 200 mg + Placebo to Etanercept
Drug: MK-3222 100 mg — MK-3222 100 mg administered SC.
  Arms: MK-3222 100 mg + Placebo to Etanercept
Drug: Placebo to MK-3222 — Matching placebo to MK-3222 administered SC.
  Arms: Placebo to MK-3222 + Etanercept 50 mg; Placebo to MK-3222 + Placebo to Etanercept
Drug: Placebo to Etanercept — Matching placebo to etanercept for subcutaneous injection.
  Arms: MK-3222 100 mg + Placebo to Etanercept; MK-3222 200 mg + Placebo to Etanercept; Placebo to MK-3222 + Placebo to Etanercept
Drug: Etanercept 50 mg — Etanercept 50 mg for subcutaneous injection.
  Arms: Placebo to MK-3222 + Etanercept 50 mg

SUMMARY:
This study is being conducted to evaluate the efficacy and safety/tolerability of SCH 900222/MK-3222 in a population of participants with moderate-to-severe plaque psoriasis.

DETAILED DESCRIPTION:
The base study consists of a screening phase of up to 4 weeks followed by a treatment period of 28 weeks, and a 20-week safety follow-up period off drug. The base study is divided into 2 sequential parts.

In Part 1 of the base study (Week 0 to Week 12), participants will be randomized to one of 4 study arms (Arm A: MK-3222 200 mg at Week 0 and Week 4 + matching placebo to etanercept twice weekly; Arm B: MK-3222 100 mg at Week 0 and Week 4 + matching placebo to etanercept twice weekly; Arm C: Matching placebo to MK-3222 at Week 0 and Week 4 + matching placebo to etanercept twice weekly; Arm D: Matching placebo to MK-3222 at Week 0 and Week 4 + etanercept 50 mg twice weekly).

In Part 2 of the base study (Week 12 to Week 28), participants in Arm A, Arm B, and Arm D will receive matching placebo to MK-3222 to maintain blinding at Week 12. Participants in Arm A and Arm B will continue to receive either MK-3222 200 mg (Arm A) or MK-3222 100 mg (Arm B) at Week 16 and Week 28 and will also receive matching placebo to etanercept once weekly through study Week 28. At study Week 12, Arm C participants will be re-randomized to receive their first dose of MK-3222 200 mg or MK-3222 100 mg, and will receive additional doses of study medication according to their re-randomized treatment assignment at Week 16 and Week 28. Participants in Arm C will also receive matching placebo to etanercept once weekly through treatment Week 28. Participants in Arm D will continue with once weekly doses of etanercept through study Week 28 in combination with matching placebo to MK-3222.

For all participants, completion of Week 28 marks completion of Part 2 and of the overall base study. Participants originally assigned to Arm D and participants who discontinue treatment prior to completing Part 2 will not be eligible to enroll in the extension. Participants that are ineligible or opt not to enter the extension study will be encouraged to complete the 20-week follow-up period.

Eligible participants that choose to enroll in the extension study will have an additional treatment period of up to 192 weeks and will be followed for an additional 20 weeks in the follow-up period. Each participant will receive MK-3222 200 mg or MK-3222 100 mg every 12 weeks up to study Week 220 according to their treatment assignment at the conclusion of Part 2 of the base study.

ELIGIBILITY:
Inclusion Criteria

* Clinical diagnosis of moderate-to-severe plaque psoriasis for at least 6 months prior to enrollment;
* Candidate for phototherapy or systemic therapy;
* Premenopausal female participants must agree to abstain from heterosexual activity or use a medically approved method of contraception or use appropriate effective contraception as per local regulations or guidelines
* For the extension study: must have completed Part 2 of the base study
* For the extension study: must have achieved at least a PASI-50 response by the end of Part 2 of the base study

Exclusion Criteria:

* Non-plaque forms of psoriasis
* Presence or history of severe psoriatic arthritis that is well-controlled on current treatment regimen
* Women of childbearing potential that are pregnant, intend to become pregnant, or are lactating
* Participant is expected to require topical therapy, phototherapy, or systemic therapy
* Presence of any infection or history of recurrent infection requiring treatment with systemic antibiotics
* Previous use of MK-3222/SCH 900222, or other interleukin-23 (IL-23)/T- helper cell 17 (Th-17) pathway inhibitors including P40, P19, and IL-17 antagonists, or etanercept
* Latex allergy or sensitivity
* Active or untreated latent tuberculosis (TB)
* For the extension study: women of child-bearing potential that are pregnant, intend to become pregnant within 6 months of completing the trial, or that are breast feeding
* For the extension study: active or uncontrolled significant organ dysfunction or clinically significant laboratory abnormalities
* For the extension study: expected to require topical treatment, phototherapy, or systemic treatment during the extension study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-09; Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants Achieving a Psoriasis Area Severity Index 75% (PASI-75) at Week 12 | Week 12
Proportion of Participants With a Physician's Global Assessment (PGA) Score of Clear or Minimal With at Least a 2 Grade Reduction From Baseline at Week 12 | Baseline, Week 12

SECONDARY OUTCOMES:
Proportion of Participants Achieving PASI-90 Response at Week 12 and 28 | Week 12, Week 28
Mean Change From Baseline in the Dermatology Life Quality Index (DLQI) at Week 12 and Week 28 | Week 12, Week 28
Proportion of Participants With a DLQI Score of 0 or 1 at Week 12 and Week 28 | Week 12, Week 28
Mean Change and Mean Percent Change from Baseline in PASI Score Over Time | Baseline, Up to Week 28
Mean Change From Baseline in the Nail Area Psoriasis Severity Index (NAPSI) at Week 12 and Week 28 | Week 12, Week 28
Number of Participants Experiencing an Adverse Event (AE) | Up to Week 28
Number of Participants Discontinuing Study Treatment Due to an AE | Up to Week 28
Proportion of Participants Achieving PASI-100 Response at Week 12 and 28 | Week 12, Week 28